CLINICAL TRIAL: NCT03324347
Title: Dog-Assisted Therapy in Dental Care Settings
Brief Title: Dog-Assisted Therapy in Dentistry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/1078 (REK)
Record Dates: First submitted 2017-10-11; First posted 2017-10-27 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2018-10

CONDITIONS: Dental Anxiety; Pediatric Dentistry; Animal Assisted Therapy
Keywords: Animal-Assisted Intervention; Dog-Assisted Intervention; Dental Care; Questionnaire; Pilot Project; Dental Clinic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapydog (Experimental): A certified therapydog (together with a certified dog-handler) will be present in the dental clinic while the child will undergo a clinical dental examination by licenced pediatric dentist.
  Interventions: Procedure: Therapydog
- No therapydog (No Intervention): No therapydog will be present in the dental clinic while the child will undergo a clinical dental examination by licenced pediatric dentist.

INTERVENTIONS:
Procedure: Therapydog — Presence of a therapydog during a clinical examination in a dental clinic
  Arms: Therapydog

SUMMARY:
Dog-assisted therapy (DAT) is used in several contexts within various areas of health care. One documented effect is that the proximity of a dog may lower anxiety in perceived stressful situations. Many individuals are afraid to visit the dentist, and someone to the extent that they need medication or anesthesia in order to complete their dental treatment. Based on the literature and own empirical observations, the investigators believe that dog-assisted therapy in connection with dental care may have a positive effect on children with dental anxiety or children that avoid dental care. It is desirable to restrict the use of drugs for these patients because of associated risk and side effects.

The purpose of this pilot study is to evaluate whether using a specially trained therapy dog can have a positive effect on children who are afraid in a dental care setting. Eligible participants (n=16) will meet twice at the dental clinic; one treatment session with a therapy dog in the dental clinic and one without. The therapy dog will be accompanied by a certified dog handler. The investigators will measure physiological variations before, during and after the treatment session. The guardian will complete validated questionnaires portraying the participant's experience of previous dental care. The participant and their guardian will also complete validated questionnaires describing their reactions from the two treatment sessions. A descriptive log for each session will be completed by the investigators.

ELIGIBILITY:
Inclusion Criteria:

* Children who are afraid of visiting the dental office / children who avoid dental treatment,
* Children who accept the presence of a dog,
* Parents or guardians who accept the presence of a dog

Exclusion Criteria:

* Children or parent/guardian that are afraid of dogs,
* Children or parent/guardian with known dog allergy,
* Children who are immunocompromised,
* Children who cannot understand or complete the patient-questionnaire

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Examination achieved; Yes or No | up to 8 weeks
  Whether the child complied or not, so that a clinical oral examination could be accomplished within 30 minutes

SECONDARY OUTCOMES:
Child satisfaction | up to 8 weeks
  The child will describe his/her feelings by marking one of 6 different emoticon-style facial expressions where number 1 illustrate the most happy face and number 6 illustrates not happy at all.
Measurement of anxiety through the CFSS-DS scale (Dental subscale of Children's Fear Survey Schedule) | up to 8 weeks
  The parent/guardian will describe the child's dental fear on a five point scale where 1 is no fear and 5 is the worst fear.
Salivary cortisol level | up to 8 weeks
  Measurement of cortisol from participant's saliva sample to assess if dog-assisted therapy (DAT) minimizes stress and anxiety
Heart rate variability | up to 8 weeks
  Heart rate will be measured to assess if dog-assisted therapy (DAT) minimizes stress and anxiety. (Biopac Systems software)
Skin conductance (Electrodermal activity) | up to 8 weeks
  Skin conductance will be measured to assess if dog-assisted therapy (DAT) minimizes stress and anxiety. (Biopac Systems software)

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Gussgard, DDS,MSc,PhD, Principal Investigator — Department of Clinical Dentistry, UiT The Arctic University of Norway
Locations (1):
- Department of Clinical Dentistry, UiT The Arctic University of Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: Undecided